CLINICAL TRIAL: NCT02636205
Title: The Use of Armeo Spring in Upper Extremity Rehabilitation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator changed. Study protocol may under go change with addition of new investigators.
Sponsor: St Mary's Hospital for Children (Other)
Responsible Party: Principal Investigator, Swetha Krishnaswamy, Occupational Therapist, St Mary's Hospital for Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-01
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Hemiplegia; Cerebral Palsy; Upper Extremity Weakness
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Armeo (Experimental): Group receiving Armeo therapy
  Interventions: Device: Armeo therapy

INTERVENTIONS:
Device: Armeo therapy — Participants will receive 18 sessionsx30 mins of ArmeoSpring therapy over 6weeks.

SUMMARY:
The purpose of this study is to evaluate the use of the Armeo®Spring Pediatric as therapy for children with hand and arm weakness. The Armeo®Spring Pediatric is a device that supports the weight of the child's arm and uses joystick that helps to play computer games. The child will be assessed before and after this therapy. Participating children with upper extremity impairments will receive therapy 3x/week for 6 weeks during 30-45 minutes sessions at progressively increasing degrees of difficulty. Each child's performance will be tracked with regard to time necessary to complete a predetermined number of trials of the activity. The standardized assessment tools that will be used are the Assisting Hand Assessment (AHA), Box & Blocks test, Jebsen Taylor hand function test, and the Pediatric Evaluation of Disability Inventory-Computer Adaptive Test (PEDI-CAT). Data will be analyzed to determine the efficacy of this training method.

DETAILED DESCRIPTION:
8. "Adverse Events" All serious adverse events will be reported to the IRB immediately, but no later than [5] days of the occurrence or receipt of notification from an outside source; the IRB can make changes to the consent form as a result of adverse events. Any such event will be reported to the IRB on the "Adverse Event Report." [See attachment.] 9. "Debriefing" Debriefing is not required because there is no deception of subjects involved or there are no alternative treatments or procedures used in a "blind" fashion.

10. "Intervention" Participants in this study are children who present with a diagnosis of upper extremity weakness or involvement secondary to various reasons. These children receive occupational, physical, and/or speech services at St Mary's Hospital for Children. The children participating in this program will be receiving their occupational therapy session with the use of the Armeo®Spring Pediatric. They will also continue to receive their regular physical and speech therapy session. Once the program is completed, they will continue to receive their regular occupation therapy sessions.

11. "Confidentiality" Data sheets will be coded with a number to represent each child. The numeric data obtained regarding timed trials will be entered into a computer which is password-protected at St. Mary's Hospital for Children in Bayside, NY. Consent forms with the child's name and parental signatures and video tape or photographic images recorded during data collection will be stored in accordance with St. Mary's Hospital for Children patient privacy policy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 -17 years.
* Arm weakness secondary to various causes.
* Armeo®Spring Pediatric fit
* Upper arm measures:155mm-235mm (7 to 9.5 inches)
* Lower arm measures: 230mm-370mm (9inches to 14 inches)
* Ability to follow instructions.

Exclusion Criteria:

* Vision deficits
* Contractures that do not allow use of system.
* Spasticity that does not allow use of system.
* Osteopenia
* Recent surgeries to the involved upper extremity.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in hand function | baseline and completion (6-8 weeks)
  Box and Blocks test
Change in hand function | baseline and completion (6-8weeks)
  Jebsen Taylor Hand Function Test
Change in bimanual hand function | baseline and completion (6-8 weeks)
  Assisting hand Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Swetha Krishnaswamy, MS OTR/L, Principal Investigator — St Mary's Hospital for Children

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- Available data/document: Study Protocol: 25014045 — http://www.ncbi.nlm.nih.gov/pubmed/25014045
- Available data/document: Study Protocol: 21261965 — http://www.ncbi.nlm.nih.gov/pubmed/?term=The+Armeo+Spring+as+training+tool+to+improve+upper+limb+functionality+in+multiple+sclerosis%3A+a+pilot+study